# Testing Financial Incentive Interventions in Dyadic-Smoker Couples NCT04832360

**Document Date: November 11, 2020** 

# UNIVERSITY OF GEORGIA CONSENT FORM SMOKING IN COUPLES

#### Researcher's Statement

You are being asked to take part in a research study sponsored by the National Cancer Institute. The information in this form will help you decide if you want to be in the study. Please ask the researcher below if there is anything that is not clear or if you need more information.

**Principal Investigator:** Dr. Michelle vanDellen

Psychology Department vandellenlab@gmail.com

- You are being asked to participate in a research study about smoking in the context of romantic relationships where both partners currently smoke. Both you and your partner must be 18 years of age or older, must be smokers, must live together, and must have internet access.
- Your involvement in the study is voluntary, and you may choose not to participate or to stop at any time without penalty or loss of benefits to which you are otherwise entitled.
- Your participation includes two 1-hour research sessions separated by three months. You have a choice to complete the two research sessions either in-person outside of the University of Georgia Psychology department or online via video conference. There will also be 10 weekly text message surveys that take less than five minutes in between the research sessions. You may also participate in an online program designed to teach about quitting smoking that consists of 4 up-to-1-hour modules that include online videos, slide presentations, and worksheets.
- The study procedures include questionnaires about your relationship, yourself, and your smoking habits; short surveys about smoking and use of quitting resources; and breathing into a machine that will read your carbon monoxide levels.
- The questionnaires and surveys will ask questions about your smoking habits, your motivation to quit, and your relationship satisfaction. This might cause discomfort to you as individuals and within your relationship. The information you provide could be embarrassing if there were a breach of confidentiality. You may also experience withdrawal if you attempt to quit smoking.
- You may benefit from the study by having access to training on smoking cessation and nicotine replacement therapy. You may also learn about yourself, your smoking behaviors, and your relationship.
- An alternative option for obtaining nicotine replacement patches/gum is to purchase these items
  from a pharmacy. An alternative option for accessing a program designed to help you quit
  smoking is to visit these websites, or search for the Beat the Pack program, which has been
  offered by the UGA College of Pharmacy:
  - o <a href="https://www.nhlbi.nih.gov/health/educational/healthdisp/pdf/tipsheets/Tips-to-Quit-Smoking.pdf">https://www.nhlbi.nih.gov/health/educational/healthdisp/pdf/tipsheets/Tips-to-Quit-Smoking.pdf</a>
  - https://smokefree.gov/tools-tips/text-programs

If you are interested in participating in the study, please read the additional information on the following pages, and feel free to ask questions at any point.

## Information about COVID-19 if you choose to participate in-person

Although the study team will attempt to reduce the risk of COVID- 19 infection during your participation, there is still a risk that you may become ill with this infection. This could lead to severe respiratory or other organ failure, and death. These complications would be more likely if you have one of the higher risk health conditions. According to the Centers for Disease Control and Prevention, people who smoke are at increased risk of severe illness from the virus that causes COVID-19.

If you choose to participate in-person, we will ask you to self-monitor for symptoms of COVID-19 and request that if you experience symptoms to cancel your scheduled session; we may reschedule at a later date. We will send you an email with a list of symptoms for you to self-monitor one week before and another email one day before your scheduled session.

There is a risk of infection if you choose to use public transportation or ride share to commute to and from the research study site. To mitigate infection risks during the study session, the research team will require you to wear a mask that fully covers your nose and mouth and maintain social distance of at least 6 feet when possible. We will also ask you to either use provided hand sanitizer and/or wash your hands before and after the study session. The research team will be wearing face masks that fully cover their nose and mouth. We will sanitize all shared devices after each participant use.

# **Study Procedures**

In this study we will ask you to complete a 1-hour Baseline Session to fill out questionnaires about your relationship, yourself, and your smoking habits. We would also like to get a reading of your current carbon monoxide levels using a breath carbon monoxide reader; this reading involves holding your breath for 15 seconds and exhaling into a handheld machine.

For 10 weeks between the Baseline and Follow-up Session, we will send you weekly text message alerts with a link to an online survey that should take no longer than five minutes to complete. Each survey will ask brief questions about your smoking and use of quitting resources during the previous week.

About 3 months after the Baseline Session, both you and your partner will be asked to participate in the Follow-up Session to answer questionnaires about your relationship, yourself, and your smoking habits and to provide a final carbon monoxide breath reading.

In order to make this study a valid one, some information about the study will be withheld from you until everyone who is participating has completed their participation. If you would like receive the additional information, we will send you an email with a link to a summary and the initial findings from the study.

#### **Risks and Discomforts**

The questionnaires might cause discomfort to you as individuals and within your relationship. Your responses will not be shared with your partner. The information you provide could be embarrassing if there

were a breach of confidentiality, and the steps we will take to minimize that are detailed below. If at any time during or after participation in this study you would like to speak with a counselor, we recommend contacting the ASPIRE Clinic at UGA (resource information will be given to you after Baseline Session and Follow-up Session). Because of the addictive properties of cigarettes, you may experience withdrawals from quitting. However, the nicotine patches or gum should help with the withdrawals if used properly.

#### **Benefits**

The biggest benefit from participating in this study is that we are offering you free resources to quit smoking (the program designed to help you quit smoking and nicotine patches/gum, which you may choose to receive). Thus, you and your partner have the potential to quit smoking from participating in this study. You may also learn about yourself, your smoking behaviors, and your relationship.

## **Participation Compensation**

After the Baseline Session and the Follow-up Session, we will ask you to fill out paperwork in order to send your participation payments to you. We will only ask you for your social security number in order to process payments for any one check that is greater than \$100. Participation payments will be sent via two checks to your home address 10-14 days after each completed session. The first check will be payment for the Baseline Session. The second check will be payment for the Follow-up Session and may include payment for completed weekly surveys and the bonus.

You will receive \$25 for completing the Baseline Session. You will receive \$25 for completing the Follow-up Session. You will receive \$1 for each weekly online survey you complete (up to \$10 for 10 weekly surveys). Participants who complete both Baseline and Follow-up Sessions and at least 8 of the 10 weekly surveys will receive a \$15 bonus. In sum, you may be compensated \$60 for participation and may receive a \$15 bonus, for a grand total of \$75. See Table 1.

Participation in this study is voluntary and you are free to refuse to participate or to withdraw from this study at any time without penalty or loss of benefits to which you are otherwise entitled. If you choose to discontinue your participation in the study, you will receive compensation for the parts of the study that you have completed. You will only receive the maximum compensation if you complete the study in its entirety. If your relationship dissolves, or if one of you wishes to withdraw, we will also terminate your partner's participation.

# **Confidentiality of Records**

If you choose to participate, your responses in this research will be confidential. Your partner will not have access to your responses. Your responses will be stored securely in the investigator's office. Following your eligibility screening, your responses are linked with an ID number, not your personal information, and the ID numbers and personal information are stored separately. Your personal information will be retained separately from your responses for up to five years after study completion. Your social security number

may be used to process your payment for this research through the University of Georgia Psychology Department's Business Department for any one check worth over \$100.

This research involves the transmission of data over the Internet. Every reasonable effort has been taken to ensure the effective use of available technology; however, confidentiality during online communication cannot be guaranteed.

Researchers will not release identifiable results of the study to anyone other than individuals working on the project without your written consent unless required by law. This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

After identifiers are removed, the information may be shared with other researchers and/or used for future studies without additional consent.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. ClinicalTrials.gov is a website that provides information about federally and privately supported clinical trials. You can search this website at any time.

# **Participant Rights**

Now, or at any time, you may discuss questions with the experimenter. You may also contact the faculty member supervising this research, Dr. Michelle vanDellen in the Psychology Department, by email at vandellenlab@gmail.com. If you have any questions about your rights as a participant, you may contact the Institutional Review Board that approved this study at 706.542.3199 or irb@uga.edu.

Please indicate your decision regarding participation in this study below:

- I agree to participate in this study. If I want a copy of this consent form for my records, I have either asked for a copy to be emailed to me from the research team or have printed this page.
- I do not agree to participate in this study.

# Below is what participation in the study looks like and the compensation you can receive.

Table 1. Study Timeline & Payment Schedule

| | Baseline Session | Optional<br>Treatment | Weekly Surveys | Follow-up Session |
|---|---|---|---|---|
| Where? | Lab | Lab | Online | Lab |
| When? | Baseline Session | ~2 weeks after<br>Baseline Session | Each week for 10<br>weeks after<br>Baseline Session | 3 months after the<br>Baseline Session |
| How<br>Long? | 1 hour or less | 1.5 hours x 4<br>meetings | Less than five<br>minutes x 10<br>surveys | 40 minutes or less |
| What? | Questionnaires and carbon monoxide reading | Training on<br>Smoking Cessation<br>(i.e., Beat the Pack) | Brief surveys about smoking behavior and use of cessation resources | Questionnaires and carbon monoxide reading |
| Payment<br>per<br>Person | \$25 | N/A | \$1 per completed<br>survey (up to \$10<br>total) | \$25 + \$15 bonus if<br>completed at least 8 of<br>10 weekly surveys and<br>both the Baseline and<br>Follow-up Sessions* |

<sup>\*</sup>Note: If you participate in both the Baseline and Follow-up Sessions and complete at least 8 of the 10 weekly surveys, you will get a \$15 bonus. Thus, the maximum amount of money to be earned for each person is \$75 (and \$150 per couple).